CLINICAL TRIAL: NCT02757066
Title: Phase II/III Clinical Trial of NPC-15 - Verification of the Efficacy for Sleep Disorders of Children With Autism Spectrum Disorders -
Brief Title: Verification of the Efficacy of NPC-15 for Sleep Disorders of Children With Autism Spectrum Disorders
Acronym: NPC-15-5
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NPC-15-5
Record Dates: First submitted 2016-04-27; First posted 2016-04-29 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Sleep Disorders; Autism Spectrum Disorder
Keywords: Melatonin; NPC-15; Sleep disorders; Autism spectrum disorders; DSM-5
MeSH Terms: conditions — Sleep Wake Disorders; Autism Spectrum Disorder | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- NPC-15 Granules Lower Dose (Experimental): NPC-15 Granules Lower Dose group which is administered 1mg melatonin
  Interventions: Drug: NPC-15 Granules Lower Dose
- NPC-15 Granules Higher Dose (Experimental): NPC-15 Granules Higher Dose group which is administered 4 mg melatonin
  Interventions: Drug: NPC-15 Granules Higher Dose
- NPC-15 Placebo Granule (Placebo Comparator): NPC-15 Placebo Granules group which is administered placebo melatonin
  Interventions: Drug: NPC-15 Placebo Granule

INTERVENTIONS:
Drug: NPC-15 Granules Lower Dose — NPC-15 granule which contains 1mg melatonin
  Other Names: Melatonin 1mg
  Arms: NPC-15 Granules Lower Dose
Drug: NPC-15 Granules Higher Dose — Melatonin granule which contains 4 mg melatonin
  Other Names: Melatonin 4mg
  Arms: NPC-15 Granules Higher Dose
Drug: NPC-15 Placebo Granule — Melatonin placebo granule which does not contains melatonin.
  Other Names: Placebo
  Arms: NPC-15 Placebo Granule

SUMMARY:
The purpose of this study is to verify the efficacy of NPC-15 (melatonin 1 mg/d or 4 mg/d) versus placebo to sleep latency with electronic sleep diaries.

DETAILED DESCRIPTION:
This study will be a multicenter, double-blind, randomized, placebo-controlled parallel group trial. The trial has five phases; the pre-screening phase, the screening phase, double-blinded treatment phase, open label treatment phase and post-treatment phase. The screening phase comprises a screening visit where subject's initial eligibility will be evaluated. During double-blinded treatment phase, patients who meet all entry criteria for the trial will be randomized into three groups, and they will be assigned NPC-15 1 mg, 4 mg or placebo before going to bed for 2 weeks. During open label treatment phase, all patients will be administered NPC-15 1 mg, 2 mg or 4 mg on the basis of their doctors' judgements.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients aged 6 to 15 years.
* Patients with "autism spectrum disorder" diagnosed by using DSM-5.
* Patients with average of daily sleep latency persisted over 30 min and the condition is continuous over 3 months
* Patients who are out-patient, not hospitalized patient.
* Signed informed consent obtained from rearer(s)/parent(s)/guardian(s) of the patient, or signed IC or informed assent obtained from the patient themselves.

Exclusion Criteria:

* Patients with at least severity in either Conceptual area, or Social area, or Practical area of intellectual disability have judged more than "severe" by using DSM-5.
* Patients who took melatonin (including supplement) in history.
* Patients who had taken Ramelteon within 4 weeks before clinical study starts.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 196 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Sleep latency with electronic sleep diary | Week 2
  Sleep latency is a common endpoint in sleep disorders. In addition, it has been used in a randomized clinical study of sleep disorders of children with neurodevelopmental disorders.

SECONDARY OUTCOMES:
Sleep latency measured by actigraphy | Week 2
  To assess the efficacy of this drug in detail
Abnormal behavior checklist Japanese version | Week 2, 9
  To assess effects of this drug on neurodevelopment disorders
Adverse events | 10 weeks
  To assess safety of this drug
Electro cardiogram | 10 weeks
  To assess safety of this drug

CONTACTS AND LOCATIONS:
Overall Officials: Yushiro Yamashita, MD, PhD, Principal Investigator — The Department of Pediatrics and Child Health Kurume University School of Medicine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yuge K, Nagamitsu S, Ishikawa Y, Hamada I, Takahashi H, Sugioka H, Yotsuya O, Mishima K, Hayashi M, Yamashita Y. Long-term melatonin treatment for the sleep problems and aberrant behaviors of children with neurodevelopmental disorders. BMC Psychiatry. 2020 Sep 10;20(1):445. doi: 10.1186/s12888-020-02847-y. PMID 32912180